CLINICAL TRIAL: NCT01954771
Title: A Prospective, Randomized, Controlled Study on Self-monitoring of Blood Glucose (SMBG) Protocols in Predicting Glucose Levels in Senior Patients With Type 2 Diabetes Mellitus (T2DM) and Coronary Artery Disease (CAD)
Brief Title: SMBG Protocols Predicting Glucose Levels in Senior Diabetes Mellitus With CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yingsheng Zhou, MD; PhD, Director of Endocrinology and Metabolism Department of Capital Medical University Affiliated Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Z131100004013044
Record Dates: First submitted 2013-09-02; First posted 2013-10-07 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
Keywords: Diabetes mellitus; Coronary artery disease; SMBG; Elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Active Comparator): Patients will receive conventional care and keep on their usual SMBG(Self-monitoring of blood glucose) methods. Additionally, each patient will also wear a CGMS(continous glucose monitoring system) device for 72h in the first week and the last week, respectively.
  Interventions: Behavioral: SMBG; Other: CGMS
- SMBG-4 Group (Active Comparator): Capillary glucose level is measured using finger stick method by 4 times (fasting plus post-meals) every other day. Additionally, each patient will also wear a CGMS device for 72h in the first week and the last week, respectively.
  Interventions: Behavioral: SMBG; Other: CGMS
- SMBG-7 Group (Active Comparator): Capillary glucose level is measured using finger stick method by 7 times (fasting, pre-meals, post-meals and bedtime altogether) every other day. Additionally, each patient will also wear a CGMS device for 72h in the first week and the last week, respectively.
  Interventions: Behavioral: SMBG; Other: CGMS

INTERVENTIONS:
Behavioral: SMBG — Control Group Patients will receive conventional care and keep on their usual SMBG methods. Additionally, each patient will also wear a CGMS device for 72h in the first week and the last week, respectively.
  SMBG-4 Group Capillary glucose level is measured using finger stick method by 4 times (fasting plus post-meals) every other day. Additionally, each patient will also wear a CGMS device for 72h in the first week and the last week, respectively.
  SMBG-7 Group Capillary glucose level is measured using finger stick method by 7 times (fasting, pre-meals, post-meals and bedtime altogether) every other day. Additionally, each patient will also wear a CGMS device for 72h in the first week and the last week, respectively.
Other: CGMS — In this study, according to the protocol, all the patients will follow their prespecified SMBG methods and periodically visit doctor, but therapies will not be adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.

SUMMARY:
Self-monitoring of blood glucose (SMBG) is a common way to assess glycemic control in diabetes management. Multiple times of blood glucose measurements by fingerstick in the same day are of tough challenge to it. The changes and variations of glucose excursion in senior diabetics with Coronary Artery Disease (CAD)involve a safety issue besides glycated hemoglobin (GHb) value. The goal of this study is to explore modified SMBG protocols for precisely monitoring and predicting glycemic excursion, variability in senior type 2 diabetics with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Clinical diagnosis of coronary artery disease
* Age ≥65 years
* The blood glucose is controlled by diets and (or) oral hypoglycemic drugs
* BMI≤28 kg/m²
* Being able to monitor and record capillary glucose value by themselves at home

Exclusion Criteria:

* Diabetic ketoacidosis (DKA)
* Acute cardiovascular events
* Anemia
* Insulin treatment
* Incapable to perform SMBG at home

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yingsheng Zhou, MD; PhD, Principal Investigator — Capital Medical University Affiliated Beijing Anzhen Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Skyler JS, Bergenstal R, Bonow RO, Buse J, Deedwania P, Gale EA, Howard BV, Kirkman MS, Kosiborod M, Reaven P, Sherwin RS; American Diabetes Association; American College of Cardiology Foundation; American Heart Association. Intensive glycemic control and the prevention of cardiovascular events: implications of the ACCORD, ADVANCE, and VA diabetes trials: a position statement of the American Diabetes Association and a scientific statement of the American College of Cardiology Foundation and the American Heart Association. Diabetes Care. 2009 Jan;32(1):187-92. doi: 10.2337/dc08-9026. Epub 2008 Dec 17. No abstract available. PMID 19092168
- [Background] Monnier L, Colette C. Glycemic variability: should we and can we prevent it? Diabetes Care. 2008 Feb;31 Suppl 2:S150-4. doi: 10.2337/dc08-s241. PMID 18227477
- [Background] Borg R, Kuenen JC, Carstensen B, Zheng H, Nathan DM, Heine RJ, Nerup J, Borch-Johnsen K, Witte DR; ADAG Study Group. HbA(1)(c) and mean blood glucose show stronger associations with cardiovascular disease risk factors than do postprandial glycaemia or glucose variability in persons with diabetes: the A1C-Derived Average Glucose (ADAG) study. Diabetologia. 2011 Jan;54(1):69-72. doi: 10.1007/s00125-010-1918-2. Epub 2010 Oct 1. PMID 20886203
- [Background] Lipska KJ, Krumholz H, Soones T, Lee SJ. Polypharmacy in the Aging Patient: A Review of Glycemic Control in Older Adults With Type 2 Diabetes. JAMA. 2016 Mar 8;315(10):1034-45. doi: 10.1001/jama.2016.0299. PMID 26954412
- [Background] Wang P, Huang R, Lu S, Xia W, Sun H, Sun J, Cai R, Wang S. HbA1c below 7% as the goal of glucose control fails to maximize the cardiovascular benefits: a meta-analysis. Cardiovasc Diabetol. 2015 Sep 22;14:124. doi: 10.1186/s12933-015-0285-1. PMID 26392171
- [Background] Munshi MN, Segal AR, Slyne C, Samur AA, Brooks KM, Horton ES. Shortfalls of the use of HbA1C-derived eAG in older adults with diabetes. Diabetes Res Clin Pract. 2015 Oct;110(1):60-65. doi: 10.1016/j.diabres.2015.07.012. Epub 2015 Aug 3. PMID 26272739
- [Background] Hoffman RM, Shah JH, Wendel CS, Duckworth WC, Adam KD, Bokhari SU, Dalton C, Murata GH; Diabetes Outcome in Veterans Study. Evaluating once- and twice-daily self-monitored blood glucose testing strategies for stable insulin-treated patients with type 2 diabetes : the diabetes outcomes in veterans study. Diabetes Care. 2002 Oct;25(10):1744-8. doi: 10.2337/diacare.25.10.1744. PMID 12351471

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Patients received conventional care and kept on their usual SMBG methods. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  SMBG
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
- SMBG-4 Group: Capillary glucose level was measured using finger stick method by 4 times (fasting plus post-meals) every other day. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  SMBG
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
- SMBG-7 Group: Capillary glucose level was measured using finger stick method by 7 times (fasting, pre-meals, post-meals and bedtime altogether) every other day. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  SMBG
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
Period: Overall Study
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Started | 29 | 32 | 28
Completed | 22 | 29 | 25
Not Completed | 7 | 3 | 3
Not completed — Missing HbA1c of end-point | 1 | 1 | 0
Not completed — Missing CGMS of end-point | 1 | 1 | 0
Not completed — Missing HbA1c and CGMS of end-point | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group | Total
Number analyzed (Participants) | 29 | 32 | 28 | 89
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.0 [66.0 to 73.0] | 70.5 [67.0 to 74.0] | 67.0 [65.0 to 70.0] | 69.0 [66.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 10 | 31
  Male | 18 | 22 | 18 | 58
Insulin secretagogues [Number; unit: participants] — include sulfonylureas and glinides
  participants
    yes | 12 | 13 | 16 | 41
    no | 17 | 19 | 12 | 48
Other Oral Anti-diabetic Drugs [Number; unit: participants]
  yes | 24 | 27 | 25 | 76
  no | 5 | 5 | 3 | 13
Statins [Number; unit: participants]
  yes | 27 | 26 | 25 | 78
  no | 2 | 6 | 3 | 11
β-blocker [Number; unit: participants]
  yes | 20 | 17 | 17 | 54
  no | 9 | 15 | 11 | 35
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 125.0 [115.0 to 136.5] | 129.0 [121.5 to 142.3] | 127.0 [116.0 to 132.5] | 128.0 [118.5 to 136.5]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 68.0 [62.0 to 73.0] | 65.5 [60.3 to 78.8] | 68.0 [60.5 to 80.0] | 67.0 [61.3 to 78.8]
Heart rate [Median (Inter-Quartile Range); unit: beats per minute] | 66.0 [59.3 to 79.0] | 72.0 [64.0 to 75.0] | 66.0 [60.0 to 71.8] | 67.0 [62.0 to 74.0]
Body mass index [Median (Inter-Quartile Range); unit: kg/m²] | 26.1 [23.3 to 28.5] | 26.1 [23.3 to 28.6] | 26.3 [23.8 to 30.2] | 26.1 [23.3 to 28.4]
Glycated hemoglobin(Normal values range from 4-6 percent) [Median (Inter-Quartile Range); unit: percent] | 7.0 [6.4 to 7.9] | 6.8 [6.5 to 7.1] | 6.8 [6.3 to 7.9] | 6.8 [6.4 to 7.5]
Hemoglobin(Normal values range from 130-175 g/L) [Median (Inter-Quartile Range); unit: g/L] | 139.0 [134.0 to 148.0] | 139.5 [121.5 to 142.3] | 143.0 [131.0 to 147.8] | 141.0 [133.0 to 148.0]
Fasting glucose(Normal values range from 3.9-6.1 mmol/L) [Median (Inter-Quartile Range); unit: mmol/L] | 7.6 [6.8 to 8.7] | 6.5 [5.7 to 8.4] | 7.5 [6.3 to 8.2] | 7.4 [6.2 to 8.4]
C-peptid(Normal values range from 0.78-5.19 ng/ml) [Median (Inter-Quartile Range); unit: ng/ml] | 1.94 [1.69 to 2.50] | 2.00 [1.30 to 2.58] | 1.87 [1.17 to 2.79] | 1.97 [1.39 to 2.56]
Insulin(Normal values range from 2.08-10.9 μU/ml) [Median (Inter-Quartile Range); unit: μU/ml] | 8.8 [6.0 to 13.0] | 9.2 [7.1 to 12.6] | 8.1 [5.1 to 15.3] | 9.0 [5.6 to 13.4]
Triglyceride(Normal values range from 0-1.7 mmol/L) [Median (Inter-Quartile Range); unit: mmol/L] | 1.35 [1.23 to 1.81] | 1.15 [0.74 to 1.86] | 1.12 [1.00 to 1.27] | 1.24 [0.79 to 1.63]
Total cholesterol(Normal values range from 3.1-5.2 mmol/L) [Median (Inter-Quartile Range); unit: mmol/L] | 3.88 [3.40 to 4.72] | 4.01 [3.34 to 4.89] | 3.46 [3.20 to 4.09] | 3.85 [3.27 to 4.48]
High density lipoprotein cholesterol(Normal values range from 1.04-1.55 mmol/L) [Median (Inter-Quartile Range); unit: mmol/L] | 1.09 [0.94 to 1.24] | 1.13 [0.98 to 1.43] | 1.12 [1.00 to 1.27] | 1.11 [0.98 to 1.28]
LDL-C (1.27-3.12 for normal; <2.59 at high risk factors; <1.80 at very high risk factors) [Median (Inter-Quartile Range); unit: mmol/L] | 2.22 [1.77 to 2.78] | 2.17 [1.72 to 2.91] | 1.85 [1.46 to 2.38] | 2.02 [1.59 to 2.68]
Blood urea nitrogen（Normal values range from 2.8-7.2 mmol/L） [Mean (Standard Deviation); unit: mmol/L] | 5.6 (1.4) | 6.2 (1.4) | 6.0 (1.4) | 5.9 (1.4)
Creatinine（Normal values range from 59-104 mmol/L for male,45-84 mmol/L for female） [Mean (Standard Deviation); unit: mmol/L] | 82.71 (15.20) | 81.65 (16.49) | 76.33 (18.87) | 80.32 (16.91)
Urinary albumin ratio(Normal values range from 0-30 mg/g) [Median (Inter-Quartile Range); unit: mg/g] | 7.59 [4.40 to 31.93] | 9.09 [4.40 to 37.57] | 8.62 [3.34 to 16.49] | 8.62 [3.84 to 23.00]
CKD-EPI -eGFR [Median (Inter-Quartile Range); unit: ml/min/1.73m²] — Chronic Kidney Disease Epidemiology Collaboration - Estimate glomerular filtration rate (CKD-EPI -eGFR)
  ml/min/1.73m² | 72.72 [66.81 to 86.66] | 80.32 [66.73 to 87.94] | 87.15 [72.93 to 92.94] | 80.81 [66.88 to 88.59]
MDRD-eGFR [Median (Inter-Quartile Range); unit: ml/min/1.73m²] — Modification of Diet in Renal Disease - Estimate glomerular filtration rate (MDRD -eGFR)
  ml/min/1.73m² | 79.39 [71.60 to 96.18] | 89.66 [75.75 to 99.80] | 93.86 [77.98 to 110.57] | 89.72 [75.54 to 100.37]

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Peak and Nadir Glucose Profiles From Continuous Glucose Monitoring System (CGMS)
Description: The peak value:>16.7mmol/L(which may precipitate ketosis),nadir:≤2.8mmol/L(Severe hypoglycemia).
Time Frame: 12 weeks
Population: 13 patients did not followed the study protocol.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Groups:
- Control Group: SMBG: Patients received conventional care and kept on their usual SMBG methods. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
- SMBG-4 Group: SMBG: Capillary glucose level was measured using finger stick method by 4 times (fasting plus post-meals) every other day. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
- SMBG-7 Group: SMBG: Capillary glucose level was measured using finger stick method by 7 times (fasting, pre-meals, post-meals and bedtime altogether) every other day. Additionally, each patient also wore a CGMS device for 72h in the first week and the last week, respectively.
  CGMS: In this study, according to the protocol, all the patients followed their prespecified SMBG methods and periodically visited doctor, but therapies were not adjusted unless they experience severe hypoglycemia or hyperglycemia episodes. The expected duration of the trial is 12 weeks.
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Number analyzed (Participants) | 29 | 32 | 28
mmol/L
  Peak at baseline | 8.86 [7.44 to 10.43] | 8.72 [7.59 to 10.22] | 8.80 [7.13 to 9.88]
  Nadir at baseline | 6.87 [5.34 to 7.65] | 6.05 [5.60 to 6.93] | 6.15 [4.95 to 7.45]
  Peak at endpoint: number analyzed (Participants) | 22 | 29 | 25
  Peak at endpoint | 8.74 [7.68 to 10.02] | 8.00 [6.34 to 8.79] | 8.68 [7.12 to 9.80]
  Nadir at endpoint: number analyzed (Participants) | 22 | 29 | 25
  Nadir at endpoint | 6.32 [5.41 to 7.59] | 6.55 [5.60 to 7.81] | 6.44 [5.89 to 8.14]

2. Secondary Outcome: The Correlation Study Between HbA1c and Glycemic Profiles of MBG (Mean Blood Glucose) From SMBG Protocols and CGMS
Description: A correlation coefficient of 0.5 is defined as large effect size.(Cohen Jacob.Statistical power analysis for the the behavioral sciences.2nd edition.Lawrence Erlbaum Associates.1988:80)
Time Frame: 12 weeks
Population: 13 patients did not followed the study protocol.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Number analyzed (Participants) | 29 | 32 | 28
mmol/L
  MBG from SMBG: number analyzed (Participants) | 22 | 29 | 25
  MBG from SMBG | 7.92 [6.99 to 8.65] | 8.00 [7.43 to 8.83] | 7.81 [7.28 to 8.61]
  MBG from CGMS at endpoint: number analyzed (Participants) | 22 | 29 | 25
  MBG from CGMS at endpoint | 7.62 [6.94 to 8.56] | 7.24 [6.64 to 8.74] | 7.76 [7.05 to 8.11]
Statistical Analysis 1: Comparison: Control Group; The correlation study between HbA1c and MBG (mean blood glucose) from SMBG measurements; Test type: Superiority or Other; p < 0.001, Correlation analysis; Correlation coefficient = 0.726
Statistical Analysis 2: Comparison: SMBG-4 Group; The correlation study between HbA1c and MBG (mean blood glucose) from SMBG measurements; Test type: Superiority or Other; p = 0.004, Correlation analysis; Correlation coefficient = 0.522
Statistical Analysis 3: Comparison: SMBG-7 Group; The correlation study between HbA1c and MBG (mean blood glucose) from SMBG measurements; Test type: Superiority or Other; p < 0.001, Correlation analysis; Correlation Coefficient = 0.784
Statistical Analysis 4: Comparison: Control Group; The correlation study between HbA1c and MBG (mean blood glucose) from CGMS measurements; Test type: Superiority or Other; p = 0.011, Correlation analysis; Correlation Coefficient = 0.533
Statistical Analysis 5: Comparison: SMBG-4 Group; The correlation study between HbA1c and MBG (mean blood glucose) from CGMS measurements; Test type: Superiority or Other; p = 0.009, Correlation analysis; Correlation Coefficient = 0.479
Statistical Analysis 6: Comparison: SMBG-7 Group; The correlation study between HbA1c and MBG (mean blood glucose) from CGMS measurements; Test type: Superiority or Other; p < 0.001, Correlation analysis; Correlation Coefficient = 0.801

3. Secondary Outcome: Number of Participants With Severe Hypoglycemia (≤50 mg/dL or 2.8mmol/L),Captured by SMBG Method and CGMS
Description: Severe hypoglycemia is defined as glucose concentration of ≤2.8mmol/L (50 mg/dL).
Time Frame: 12 weeks
Population: 13 patients did not followed the study protocol.
Measure: Number; unit: participants
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Number analyzed (Participants) | 29 | 32 | 28
participants
  Baseline CGMS | 4 | 3 | 7
  End-point CGMS: number analyzed (Participants) | 22 | 29 | 25
  End-point CGMS | 3 | 1 | 3
  SMBG | 1 | 0 | 1

4. Secondary Outcome: HbA1c(%) at Endpoint
Time Frame: 12 weeks
Population: 13 patients did not followed the study protocol.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Number analyzed (Participants) | 22 | 29 | 25
percentage | 6.9 [6.2 to 7.2] | 6.7 [6.1 to 7.0] | 6.6 [6.4 to 7.3]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Events reported according to description in study protocol.
Arm/Group | Control Group | SMBG-4 Group | SMBG-7 Group
Serious Adverse Events (participants affected / at risk) | 7/29 | 4/32 | 7/28
Other Adverse Events (participants affected / at risk) | 16/29 | 20/32 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=29) | SMBG-4 Group (N=32) | SMBG-7 Group (N=28)
Severe hypoglycemia (≤2.8mmol/L) (Endocrine disorders) | 7 (7) | 4 (4) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=29) | SMBG-4 Group (N=32) | SMBG-7 Group (N=28)
Hemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (≤3.9mmol/L) (Endocrine disorders) | 16 (16) | 20 (20) | 19 (19)
Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This clinical trial population may not be representative of all patients. Because patients missed clinic visits in three months by reason of vacation tour, or complained about frequent blood samplings, 14.6% of all did not follow the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less